CLINICAL TRIAL: NCT06423079
Title: Complex Intaocular Lens-Bag Fixation With Siepser's Scleral Sliding Knots
Brief Title: Scleral Fixation for Intraocular Lens-Bag Dislocation
Status: Completed | Type: Observational
Sponsor: University of Naples (Other)
Responsible Party: Principal Investigator, Luca D'Andrea, Prinicipal investigator, University of Naples
Other Study IDs: Siep_001
Record Dates: First submitted 2024-05-15; First posted 2024-05-21 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Pseudoexfoliation Syndrome
MeSH Terms: conditions — Exfoliation Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- IOL-Bag Dislocation patients: Patients affected by pseudoexfoliation syndrome, with inferior dislocation of the bag-IOL complex.
  Interventions: Procedure: Siepser knots

INTERVENTIONS:
Procedure: Siepser knots — Surgical intervention involved creating a superior service keratotomy and using introflective sutures for IOL fixation

SUMMARY:
Novel introflective sutures offer a minimally invasive approach for stable fixation of dislocated bag-IOL complexes, preserving visual acuity and reducing corneal complications in patients with pseudoexfoliation syndrome.

DETAILED DESCRIPTION:
To assess the one-month outcomes of visual performance and positional stability of capsule-fixated intraocular lenses (IOLs) in patients with IOL-Bag complex dislocation. Patients with intraoperative complications or prior posterior capsule Nd-YAG laser were excluded. Surgical intervention involved creating a superior service keratotomy and using introflective sutures for IOL fixation. Best Corrected Visual acuity (BCVA), endothelial cell counts, and tonometry were assessed at multiple postoperative time points. We also evaluated the mean spherical equivalent (SE), and the residual cylinder and sphere at each follow-up.

ELIGIBILITY:
Inclusion Criteria:

* patients affected by pseudoexfoliation syndrome, with inferior dislocation of the bag-IOL complex

Exclusion Criteria:

* patients who underwent intraoperative complications,
* dislocation in the vitreous chamber of the bag-IOL complex,
* patients who had already undergone posterior capsule Nd-YAG laser

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients affected by pseudoexfoliation syndrome, with inferior dislocation of the bag-IOL complex after cataract surgery.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2017-05-10 (Actual); Primary Completion 2019-05-10 (Actual); Study Completion 2022-05-10 (Actual)

PRIMARY OUTCOMES:
Best corrected visual acuity | 1 year
  to evaluate the best corrected visual acuity after the surgery

SECONDARY OUTCOMES:
Endothelial cells count | 1 year
  to evaluate the Endothelial cells count after the surgery

CONTACTS AND LOCATIONS:
Locations (1):
- University of Naples Federico II, Naples, Italy

IPD SHARING:
Plan to Share IPD: Yes
all collected IPD
Time Frame: 5 years
Access Criteria: available on request
URL: https://guides.lib.umich.edu/datamanagement/clinicaltrials

REFERENCES:
- [Derived] Furgiuele D, Giunta P, Rinaldi M, D'Andrea L, Costagliola C. Innovative approach to IOL-bag complex fixation with Siepser's scleral sliding knots in pseudoexfoliation syndrome. Sci Rep. 2025 Aug 5;15(1):28522. doi: 10.1038/s41598-025-10542-9. PMID 40764517